CLINICAL TRIAL: NCT01249248
Title: PD2i Analysis of Heart Rate Variability in Competitive Sports
Acronym: PACA
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Vicor Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, James Hughes, Professor, University of Mississippi Medical Center
Other Study IDs: 2010-0158
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Autonomic Dysfunction
Keywords: Heart rate variability; Autonomic dysfunction; Exercise; Sports; Competition; Athletes
MeSH Terms: conditions — Primary Dysautonomias; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Male basketball players
  Interventions: Device: PD2i Analyzer
- Female basketball players
  Interventions: Device: PD2i Analyzer
- Baseball players
  Interventions: Device: PD2i Analyzer
- Softball players
  Interventions: Device: PD2i Analyzer
- Football players
  Interventions: Device: PD2i Analyzer
- Female vollyball players
  Interventions: Device: PD2i Analyzer
- Male soccer players
  Interventions: Device: PD2i Analyzer
- Female soccer players
  Interventions: Device: PD2i Analyzer

INTERVENTIONS:
Device: PD2i Analyzer — Analysis of heart rate variability from a standard digital ECG for 6-12 minutes

SUMMARY:
This is a double blind observational analysis of changes in heart rate variability using PD2i analyser in competitive athletes during strenuous exercise and competition.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, as determined by birth date given on participation form.
* Actively involved in competitive athletics
* Able to give informed consent

Exclusion Criteria:

* Any known prior autonomic dysfunction
* History of seizures or taking anti-seizure medication
* Known learning disability or attention deficit disorder
* Chronic heart conditions such as arrhythmias or valvular disease
* History of diabetes mellitus
* Taking any prescription stimulants such as Ritalin, Focalin, etc.
* Use of any performance-enhancing drugs
* Any deviation from normal found on the pre-participation physical exam such as the presence of a murmur or hypertension.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: College athletes on competitive teams.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in PD2i following strenuous exercise bout of 45 minutes | Baseline at zero minutes and within 60 minutes of completion of strenuous exercise bout.
  PD2i analysis of HRV measured before and after strenuous exercise in each sport. The change from baseline will be correlated to return to resting heart rate.

SECONDARY OUTCOMES:
Change in PD2i following an injury during competitive sports. | Baseline PD2i at zero and within 60 minutes of cessation of exercise bout.
  If an athlete participating in the research sustains an injury the PD2i analysis will be obtained and correlated to the baseline analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Steve A Watts, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States